CLINICAL TRIAL: NCT01308008
Title: Home Program to Enhance Mobility in Older Veteran Diabetics
Brief Title: Home Exercise to Enhance Mobility for Older Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E7547-R
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Type 2 Diabetes Mellitus; Mobility Limitation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Mobility Limitation | interventions — Exercise; Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional exercise- home physical activity (Experimental): On-site personal trainer-based functional aerobic program followed by home intervention consisting of functional exercise training and enhanced physical activity with telephonic behavioral support
  Interventions: Behavioral: home exercise/physical activity (PA) enhancement program with behavioral support
- Flex and tone- home health education (Active Comparator): Initial on-site flex and toning program continued on follow-up along with health education
  Interventions: Behavioral: flex and toning health education program

INTERVENTIONS:
Behavioral: home exercise/physical activity (PA) enhancement program with behavioral support — Initial on-site personal trainer-based functional aerobic program followed by home intervention consisting of functional exercise training and enhanced physical activity with nurse telephonic behavioral support
  Arms: Functional exercise- home physical activity
Behavioral: flex and toning health education program — Initial flex and toning program continued on follow-up along with health education
  Arms: Flex and tone- home health education

SUMMARY:
The goal of the proposed research is to test whether a long-term exercise program in sedentary Veterans with diabetes will produce sustained improvement in mobility performance and physical activity. In this proposed research, 240 sedentary older adult diabetics (aged 60 and over) will be randomly allocated into a customized, primarily home-based, functionally-oriented exercise program with nurse support intervention (I) group versus a flexibility and toning, health education control (C) group, and test outcomes in functional mobility and physical activity at 4 weeks, 6 months and one year. This research can lead to an exercise/PA enhancement program that can coordinate with VA outreach programs, targeting older Veterans who are not in the immediate vicinity of a major VA site. Ultimately, this should create a model to which physicians and other providers could refer comorbid diabetes patients.

DETAILED DESCRIPTION:
The goal of the proposed research is to test whether a long-term exercise program in sedentary Veterans with diabetes will produce sustained improvement in mobility performance and physical activity. To facilitate adherence to a long-term program, the investigators plan an individualized, home exercise/physical activity (PA) enhancement program with behavioral support. The rationale for this program is based on: 1) the feasibility of a previously funded VA RR&D controlled trial (led by the present research team) in sedentary older adults with diabetes that improved mobility performance, specifically usual gait speed; 2) the need for longer term and functionally-relevant interventions (specifically mobility-oriented) for older adult diabetics; 3) the potential to use telephonic nurse support to assist in overcoming barriers to exercise and in dealing with intercurrent illness, factors that are key in this comorbid patient group; and 4) the potential to increase the focus on objectively measured physical activity. In this proposed research, 240 sedentary older adult diabetics (aged 60 and over) will be randomly allocated into a customized, primarily home-based, functionally-oriented exercise program with nurse support intervention (I) group versus a flexibility and toning, health education control (C) group, and test outcomes in functional mobility and physical activity at 4 weeks, 6 months and one year.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* Type 2 Diabetes
* No medical contraindications to exercise

Exclusion Criteria:

* Enrolled in intensive exercise program
* Unable to cooperate with protocol (e.g. cognitive impairment)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2011-11; Primary Completion 2016-05 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Alexander, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Ann Arbor, Michigan and surrounding communities. Recruitment relied primarily on media advertisement, community outreach and mailings to patients with diabetes treated at the Veterans Affairs Ann Arbor Healthcare System (VAAAHS) and the University of Michigan (UM), both of which provided IRB approval.
Pre-assignment Details: Withdrawal after Screening, prior to Baseline: N=5
Groups:
- Functional Exercise- Home Physical Activity: Initial on-site personal trainer-based functional aerobic program followed by home intervention consisting of functional exercise training and enhanced physical activity with nurse telephonic behavioral support
  home exercise/physical activity (PA) enhancement program with behavioral support: Initial on-site personal trainer-based functional aerobic program followed by home intervention consisting of functional exercise training and enhanced physical activity with nurse telephonic behavioral support
Period: 4 Weeks
Arm/Group | Functional Exercise- Home Physical Activity | Flex and Tone- Home Health Education
Started | 71 | 73
Completed | 62 | 71
Not Completed | 9 | 2
Not completed — Illness, disinterest, time | 9 | 2
Period: 6 Months
Arm/Group | Functional Exercise- Home Physical Activity | Flex and Tone- Home Health Education
Started | 62 | 71
Completed | 54 | 62
Not Completed | 8 | 9
Period: 12 Months
Arm/Group | Functional Exercise- Home Physical Activity | Flex and Tone- Home Health Education
Started | 54 | 62
Completed | 46 | 58
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Functional Exercise- Home Physical Activity | Flex and Tone- Home Health Education | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 71 | 73 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69 (6) | 70 (6) | 70 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 49 | 47 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 54 | 58 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Comfortable gait speed [Mean (Standard Deviation); unit: meters per second] — Gait velocity over 6 meters
  meters per second | 1.1 (0.2) | 1.1 (0.2) | 1.1 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Comfortable Gait Speed
Description: Gait velocity over 6 meters
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Functional Exercise- Home Physical Activity | Flex and Tone- Home Health Education
Number analyzed (Participants) | 71 | 73
meters per second | 1.2 (0.2) | 1.2 (0.2)
Statistical Analysis 1: Comparison: Functional Exercise- Home Physical Activity vs Flex and Tone- Home Health Education; Test type: Superiority; p = 0.16, Regression, Logistic; coefficient = 0.05, 95% CI 2-sided [-0.02 to 0.13]

2. Primary Outcome: Six Minute Walk Distance
Description: Walk distance covered in feet over 6 minutes
Time Frame: one year
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Functional Exercise- Home Physical Activity | Flex and Tone- Home Health Education
Number analyzed (Participants) | 71 | 73
feet | 1307 (234) | 1271 (275)
Statistical Analysis 1: Comparison: Functional Exercise- Home Physical Activity vs Flex and Tone- Home Health Education; Test type: Superiority; p = 0.17, Regression, Logistic; coefficient = 34.0, 95% CI 2-sided [-15 to 83]

3. Secondary Outcome: Physical Activity
Description: Average physical activity counts per waking minute
Time Frame: one year
Measure: Mean (Standard Deviation); unit: counts per minute
Arm/Group | Functional Exercise- Home Physical Activity | Flex and Tone- Home Health Education
Number analyzed (Participants) | 71 | 73
counts per minute | 170 (89) | 141 (66)
Statistical Analysis 1: Comparison: Functional Exercise- Home Physical Activity vs Flex and Tone- Home Health Education; Test type: Superiority; p = 0.5, Regression, Logistic; coefficient = -8.7, 95% CI 2-sided [-35 to 17]

ADVERSE EVENTS:
Groups:
- Functional Exercise- Home Physical Activity: Functional exercise- home physical activity
- Flex and Tone- Home Health Education: Flex and tone- health education
Arm/Group | Functional Exercise- Home Physical Activity | Flex and Tone- Home Health Education
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/73
Serious Adverse Events (participants affected / at risk) | 3/71 | 3/73
Other Adverse Events (participants affected / at risk) | 0/71 | 2/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Exercise- Home Physical Activity (N=71) | Flex and Tone- Home Health Education (N=73)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Partial achilles tendon tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to training (s/p fall off bike)
Colonic polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Exercise- Home Physical Activity (N=71) | Flex and Tone- Home Health Education (N=73)
Baker's cyst drainage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hand pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — post hand grip testing

LIMITATIONS AND CAVEATS:
Study completed with depletion of funds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No